CLINICAL TRIAL: NCT04699877
Title: A Phase 1 Open-label Study to Investigate the Effect of Severe Renal Impairment on the Pharmacokinetics, Safety and Tolerability of Gilteritinib Compared to Healthy Participants With Normal Renal Function
Brief Title: A Study to Investigate the Effect of Severe Renal Impairment on Gilteritinib Compared to Healthy Participants With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2215-CL-0114; 2020-003993-32 (EudraCT Number)
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Renal Impaired; Gilteritinib; Normal Renal Function; Pharmacokinetics of ASP2215
Keywords: Gilteritinib
MeSH Terms: interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gilteritinib (Severe Renal Impairment) (Experimental): Participants with severe renal impairment received a single oral dose of 20 milligrams (mg) of gilteritinib on day 1, under fasting conditions.
  Interventions: Drug: Gilteritinib
- Gilteritinib (Normal Renal Function) (Experimental): Participants with normal renal function received a single oral dose of 20 mg of gilteritinib on day 1, under fasting conditions.
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — Oral
  Other Names: ASP2215; XOSPATA®

SUMMARY:
The purpose of the study was to evaluate the pharmacokinetics of a single oral dose of gilteritinib in male and female participants with severe renal impairment compared to healthy male and female participants with normal renal function. This study also evaluated safety and tolerability of a single oral dose of gilteritinib in male and female participants with severe renal impairment and healthy male and female participants with normal renal function. Part 2 of the study (mild and moderate renal impairment) was not conducted based on the final pharmacokinetic findings from part 1 (severe renal impairment).

DETAILED DESCRIPTION:
This study was comprised of participants with severe renal impairment and normal renal function. Participants were residential for a single period of 14 days/13 nights. Participants were discharged from the clinical unit on day 14 on the condition that all required assessments had been performed and that there were no medical reasons for a longer stay in the clinical unit.

ELIGIBILITY:
Inclusion Criteria:

Participant is eligible for participation in the study if all of the following apply:

* Participant has body mass index (BMI) range of 18.5 to 40.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female participant is not pregnant and the following condition apply: Not a woman of childbearing potential (WOCBP)
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 120 days after Investigational Product (IP) administration.
* Male participant must not donate sperm during the treatment period and for 120 days after investigational product (IP) administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 120 days after IP administration.
* Participant has renal function defined by estimated glomerular filtration rate (eGFR) using modification of diet in renal disease (MDRD) formula:

  * Normal renal function with eGFR ≥ 90 mL/min per 1.73 m^2, or
  * Mild renal impairment with eGFR 60 to <90 mL/min per 1.73 m^2, or
  * Moderate renal impairment with eGFR 30 to <60 mL/min per 1.73 m^2, or
  * Severe renal impairment as defined by the National Kidney Foundation and by eGFR <30 mL/min per 1.73 m^2 and not on hemodialysis (preferably not higher than 20 mL/min per 1.73 m^2, with at least 50% of participants required to have eGFR ≤ 20 mL/min per 1.73 m^2).
* Participant has adequate venous access to allow collection of study-related samples.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

Participant will be excluded from participation in the study if any of the following apply:

* Participant has received any investigational therapy within 28 days or 7 half-lives, whichever is longer, prior to day -1.
* Participant has any condition which makes the participant unsuitable for study participation.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Participant has a known or suspected hypersensitivity to gilteritinib or any components of the formulation used.
* Participant has had previous exposure with gilteritinib.
* Participant has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and total bilirubin [TBL]) ≥ 1.5 × upper limit of normal on day -1. In such a case, the assessment may be repeated once.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to IP administration.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF) of > 450 msec (for male and female participants) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate 12-lead electrocardiogram (ECG) may be taken.
* Participant has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to day -1.
* Participant has a history of consuming > 14 units for male participants or > 7 units for female participants of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism 3 months prior to screening or drug/chemical/ substance abuse within 1 year prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* Participant has used any inducer of cytochrome P450 (CYP)3A metabolism (e.g., St. John's Wort, barbiturates and rifampin) in the 3 months prior to day -1.
* Participant has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Participant has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease or a family history of long QT syndrome.
* Participant has a positive serology test for hepatitis A virus immunoglobulin M antibodies, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening. Participants with isolated hepatitis B core antibody (with negative hepatitis B surface antigen and negative hepatitis B surface antibody) may be eligible if hepatitis B DNA or hepatitis C RNA is undetectable.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.
* Participant who has received any of the following drugs/products within 2 weeks prior to IP administration:

  * Strong or moderate CYP3A inhibitors (e.g., grapefruit, Seville oranges, ketoconazole or fluconazole)
  * Strong or moderate inhibitors and all inducers of P-glycoprotein
  * Substrates of multidrug and toxin extrusion 1
  * Drugs that target serotonin 5-hydroxytryptamine receptor 1 or 5-hydroxytryptamine receptor 2B
* Participant has a positive result for SARS-CoV-2 polymerase chain reaction (PCR) test during screening.
* Participant has clinical signs and symptoms consistent with COVID-19 infection, e.g., fever, dry cough, dyspnea, sore throat, muscle or body aches and gastrointestinal symptoms or confirmed infection by appropriate SARS-CoV-2 PCR test within the 4 weeks prior to screening.

Additional criteria for participants with mild, moderate and severe renal impairment:

* Participant who has a history of any clinically significant illness (other than renal disease and conditions related to renal disease, such as stable diabetes and stable hypertension), medical condition or laboratory abnormality within 3 months prior to screening which precludes the participant from study participation.
* Participant has a mean pulse rate < 40 or > 90 bpm; mean systolic blood pressure (SBP) < 90 or > 160 mmHg; mean diastolic blood pressure (DBP) < 50 or > 100 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse rate will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant who has had a change in dose regimen of medically required medication(s) in the 2 weeks prior to IP administration (permitted concomitant medications) and/or participant for whom dose changes are likely to occur during the study (minor dose changes are allowed in agreement with the sponsor) and/or participant has used nonpermitted concomitant medication(s) (including, but not limited to vitamins, hormonal contraceptives and natural and herbal remedies) in the 3 weeks prior IP administration, except for topical dermatological products (including corticosteroid products) and hormone replacement therapy (HRT).
* Participant who requires or is likely to require any new concomitant medications during the course of the study.
* Participant who has a renal disease secondary to malignancy.
* Participant who has a fluctuating or rapidly deteriorating renal function within 4 weeks prior to IP administration, as indicated by strongly varying or worsening clinical and/or laboratory signs of renal impairment within the screening period.
* Participant has a hemoglobin result of < 8.5 g/dL.
* Participant has a functioning kidney transplant.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids,cocaine and/or opiates) at screening or on day -1, unless the positive result is due to an approved prescription medication.

Additional criteria for healthy participants with normal renal function:

* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has any clinically significant abnormality following the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* Participant has a mean pulse rate < 45 or > 90 bpm; mean SBP > 150 mmHg; mean DBP > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse rate will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has used any prescribed or nonprescribed drugs (including, but not limited to vitamins, hormonal contraceptives and natural and herbal remedies) in the 2 weeks prior to IP administration, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products (including corticosteroid products) and HRT.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on day -1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of gilteritinib in plasma: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Predose on day 1 and at the following postdose time points on 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24,48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312 hour(s) and at the end of study (maximum: day 23)
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity was derived from the plasma samples.
PK of gilteritinib in plasma: Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Predose on day 1 and at the following postdose time points on 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24,48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312 hour(s) and at the end of study (maximum: day 23)
  Area under the concentration-time curve from the time of dosing to the last measurable concentration was derived from the plasma samples.
PK of gilteritinib in plasma: Maximum concentration (Cmax) | Predose on day 1 and at the following postdose time points on 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24,48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312 hour(s) and at the end of study (maximum: day 23)
  Maximum plasma concentration of gilteritinib was derived from the plasma samples.
PK of gilteritinib in plasma: Apparent clearance (CL/F) | Predose on day 1 and at the following postdose time points on 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24,48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312 hour(s) and at the end of study (maximum: day 23)
  CL/F derived from plasma samples.
Pk of gilteritinib in plasma: Area under the concentration-time curve from the time of dosing extrapolated to the time infinity (unbound)(AUCinf,u) | Predose on day 1 and at the following postdose time points on 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24,48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312 hour(s) and at the end of study (maximum: day 23)
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity (unbound) was derived from plasma samples.
PK of gilteritinib in plasma: Area under the concentration-time curve from the time of dosing to the last measurable concentration (unbound) (AUClast, u) | Predose on day 1 and at the following postdose time points on 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24,48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312 hour(s) and at the end of study (maximum: day 23)
  Area under the concentration-time curve from the time of dosing to the last measurable concentration (unbound) was derived from plasma samples.
PK of gilteritinib in plasma: Maximum concentration (unbound) (Cmax,u) | Predose on day 1 and at the following postdose time points on 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24,48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312 hour(s) and at the end of study (maximum: day 23)
  Maximum concentration of gilteritinib (unbound) was derived from plasma samples.

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to Day 23
  An AE is any untoward medical occurrence in a participant administered a study drug, which does not necessarily have to have a causal relationship with this treatment. It can, therefore, be any unfavorable and unintended sign, symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product whether considered related to the medicinal product. Treatment Emergent Adverse Event defined as an AE observed after starting administration of the study drug till 23 days.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- United States (3):
  - National Institute of Clinical Research, Garden Grove, California
  - Orange County Research Institute, Tustin, California
  - Orlando Clinical Research Center, Orlando, Florida
- Site BG35901, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.